CLINICAL TRIAL: NCT06285825
Title: A Pilot Study of Emapalumab for the Treatment of CAR T-Cell Therapy-Associated Prolonged Cytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0864; NCI-2024-01736 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cytopenia
MeSH Terms: conditions — Cytopenia | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental): If you are found to be eligible to take part in this research study, you will be assigned to 1 of 2 dose levels of emapalumab, based on when you enroll on the study. Up to 16 participants will receive each dose level of the study drug.
  * The first group of 5 participants will be enrolled at the lower dose level.
  * Depending on the safety data seen in this first group, the next 11 participants will be enrolled at the lower dose.
  * After reviewing the early safety data from that first group of 16 participants, the study team will enroll the next 5 participants at the higher dose level and be checked for serious side effects.
  * Depending on the safety information from the first 5 participants in the higher dose level group, the other 11 will then be enrolled.
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Given by Infusion

SUMMARY:
To look at the safety and effectiveness of emapalumab for the treatment of prolonged severe cytopenia in participants with LBCL who receive CART.

DETAILED DESCRIPTION:
Primary Objectives:

- To evaluate the efficacy of emapalumab for the treatment of prolonged severe cytopenia in participants with LBCL who receive CART.

Secondary Objectives:

- To evaluate safety and tolerability of emapalumab for the treatment of prolonged severe cytopenia in participants with LBCL who receive CART.

Exploratory Objective:

- To investigate biomarkers of response and resistance to emapalumab for the treatment of prolonged severe cytopenia in participants with LBCL who receive CART.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be considered for inclusion in this study if they meet the following criteria based on tests obtained less than 4 weeks from first dose:

1. Relapsed or refractory FL (grade 1, 2, 3a and 3b), MCL, DLBCL, PMBCL, tFL, or HGBCL
2. Received standard of care therapy with axi-cel, tisa-cel or liso-cel
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. Either in remission after CART and/or with refractory/progressive disease not requiring urgent treatment in the opinion of the treating physician
6. Grade 3-4 cytopenia defined as either absolute neutrophil count of < 1.0x109/L, or platelet count < 50x109/L or haemoglobin< 8 g/dL starting or persisting between day 30 and day 90 after CART
7. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 30 mL/min
8. Serum alanine transaminase (ALT) / aspartate transaminase (AST) ≤ 2.5 upper limit of normal (ULN), independently from etiology
9. Total bilirubin ≤1.5 mg/dL, or ≤ 3 UNLin participants with Gilbert's syndrome.
10. Baseline oxygen saturation > 92% on room air 11 Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)

12. Participant will be willing to undergo a bone marrow biopsy before and at the end of each cycle, and at time of severe cytopenia recurrence; archived samples can be accepted during the screening period in absence of intercurrent treatment 13. The effects of emapalumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for up to 6 months after the administration of emapalumab (whichever is administered last). (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the participants presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of emapalumab administration.

  14. Ability to understand and the willingness to sign a written informed consent document.

  15. Participant will need to test for latent tuberculosis infections using the purified protein derivative (PPD) or IFNƒÁ release assay and will be evaluated for tuberculosis risk factors within 3 months from initiation of treatment. We will administer tuberculosis prophylaxis to participants at risk for tuberculosis, or known to have a positive PPD test result, or positive IFNƒÁ release assay.

Exclusion Criteria:

Participants will be ineligible for this study if they meet the following criteria:

1. History of malignancy other than nonmelanoma skin cancer or localized carcinoma (e.g., cervix, bladder, breast, prostate) unless disease free for at least 3 years.
2. History of Richter's transformation of chronic lymphocytic leukemia (CLL)
3. Presence of grade 3-4 cytopenia before initiation of lymphodepleting chemotherapy for CART
4. Grade 3-4 cytopenia due to use of experimental non-commercially available CART product
5. Bone marrow evidence of LBCL, hypersplenism, HLH, or a second malignancy (e.g., MDS) that could be contributing to cytopenia, with no alternative, identifiable potential cause for the cytopenia.
6. Relapsed or progressive disease requiring immediate initiation of anti-lymphoma treatment
7. Known presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management, including leishmania infection. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Principal investigator.
8. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). A history of HIV, hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing. For participants with a history of Hepatitis B or C, standard of care monitoring for viral reactivation will be conducted. Subjects with a history of Hepatitis B will be required to undergo hepatitis B reactivation prophylaxis unless contraindicated.
9. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrolment
10. History of primary immunodeficiency
11. History of symptomatic deep vein thrombosis or symptomatic pulmonary embolism within 1 month of enrolment considered significant in the opinion of the principal investigator
12. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment in the investigator's opinion
13. History of severe immediate hypersensitivity reaction to any of the agents used in this study, including E coli-derived proteins.
14. Receipt of BCG vaccine within 12 weeks prior screening or receipt of a live or attenuated (other than BCG) vaccine within 4 weeks prior to screening
15. Women of child-bearing potential who are pregnant or breastfeeding.
16. Women of child-bearing potential and men with partners who are of child-bearing potential who are not willing to practice birth control as noted in section 4.1 from the time of consent through 6 months after the completion of emapalumab.
17. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participationTrial Treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2028-08-22 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Strati, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org